CLINICAL TRIAL: NCT06032689
Title: Two-Years Clinical Performance of Bulk-Fill High Viscosity Ormocer Versus Methacrylate-Based Resin Composite Restorative Systems: The Effect of Bulk-Fill Low-viscosity Resin Composite Liners in Class II Restorations.
Brief Title: A 2-year Clinical Impact of Bulk-fill Low-viscosity Resin Composite Liners in Class II Restorations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M 11120520
Record Dates: First submitted 2023-08-02; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dental Caries Class II

STUDY DESIGN:
Intervention Model Description: participants had at least four class II cavities in a split-mouth design and randomly each cavity was restored using one of four strategies( groups applied)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Xtra-fill (Active Comparator): Bulk-fill high-viscosity methacrylate-based resin composites.
  Interventions: Combination Product: Xtra-fill
- X-base (Active Comparator): Bulk-fill low-viscosity methacrylate-based resin composites.
  Interventions: Combination Product: x-base
- Admira fusion x-tra (Active Comparator): Bulk-fill high-viscosity ormocer-based resin composites.
  Interventions: Combination Product: Admira fusion x-tra
- Admira fusion x-base (Active Comparator): Bulk-fill low-viscosity ormocer-based resin composites.
  Interventions: Combination Product: Admira fusion x-base

INTERVENTIONS:
Combination Product: Xtra-fill — the material was placed in bulk.
  Arms: Xtra-fill
Combination Product: x-base — The x-base liner was placed and then veneered with Xtra-fill.
  Arms: X-base
Combination Product: Admira fusion x-tra — bulk placement of the restoration Admira fusion -xtra.
  Arms: Admira fusion x-tra
Combination Product: Admira fusion x-base — Admira fusion x-base liner was used and then veneered by Admira fusion x-tra.
  Arms: Admira fusion x-base

SUMMARY:
This randomized clinical trial evaluated the clinical performance of class II resin composite restorations using bulk-fill high-viscosity ormocer versus methacrylate-based with or without a thin layer of bulk-fill low-viscosity (flowable) resin composite liners (BLRC) over 2 years. The null hypotheses in the study were as follows: (1) Different types of matrix structures (ormocer vs. methacrylate) have no effect on the marginal integrity of restorations; (2) A layer of bulk-fill resin compo-site liner of the same category would not affect the marginal or internal adaptation of restorations.

DETAILED DESCRIPTION:
The study was designed following the Consolidated Standards of Reporting Trials (CONSORT) statement. approvement by the local ethics committee of Mansoura University code register was taken code M 11120520. The patients were selected as they searched for treatment in the Conservative Dentistry Department outpatient clinic, in the Faculty of Dentistry, Mansoura University. A group of 30 patients 21 Females and 9 males was chosen from among 92 participants after careful consideration of the inclusion and exclusion criteria. The sample size estimate was made based on the clinical success rate of posterior class II composite restorations observed in a prior study (97.5% at 24 months). The sample size needed per group was 23 teeth using a significance level of 0.05, power of 80%, and equivalency limit of 15%. A total of 30 patients were chosen, for a total of 120 restorations (30 for each group) after taking potential dropouts into account. To ensure adherence of the participants to the study, all volunteers underwent complete dental treatment and periodic follow-ups. The volunteers were contacted by telephone, WhatsApp message, Facebook, and e-mail for the assessments. Four attempts, including visits to the schools, were made to contact a volunteer before he/she was considered a "loss." both participants and examiners were blind to the interventions. An inter-examiner and intra-examiner agreement of at least 90% was requested before the beginning of the evaluation. Clinical evaluation was performed one week after finishing and polishing (baseline), after 6 months, 12 months, 18 months, and 24 months using the World Dental Federation (FDI) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients having at least 4 posterior teeth with moderate occlusal-proximal carious lesions.
* Patients ranging in age from 18 to 30 years.
* patients with normal occlusion.

Exclusion Criteria:

General exclusion criteria:

* Patients having severe chronic periodontitis.
* Patients with orthodontic appliances.
* Abnormal occlusion, parafunctional habits.
* Allergy to any of the materials used in the study. Specific teeth exclusion criteria
* Teeth with irreversible pulpitis or non-vital.
* Fractured or cracked teeth.
* Previously restored teeth.
* Cavities with isthmus larger than intercuspal distance.
* Teeth with deep sub-gingival cavity margins.

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
clinical performance | two years
  FDI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sa Mahmoud, professor, Principal Investigator — Operative Dentistry
Locations (1):
- Mansoura U, Al Mansurah, Mansoura, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT06032689/Prot_SAP_000.pdf